CLINICAL TRIAL: NCT03177135
Title: PROOF OF AMNIOSENSE BLUE IN HOME USAGE AND AS A HOSPITAL STANDARD OF CARE FOR AMNIOTIC FLUID LEAK DETECTION
Brief Title: PROOF OF AMNIOSENSE BLUE IN HOME USAGE AND HOSPITAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Common Sense (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: F-7-32.3-1
Record Dates: First submitted 2017-05-28; First posted 2017-06-06 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-05

CONDITIONS: Amniotic Problems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AmnioSense diagnostic pantyliner (Experimental): AmnioSense diagnostic pantyliner of amniotic fluid compared with standard clinical diagnosis methods
  Interventions: Device: AmnioSense

INTERVENTIONS:
Device: AmnioSense — A diagnostic pantyliner for detection of amniotic fluid leaks compared with standard clinical diagnosis.

SUMMARY:
This is a Prospective study to demonstrate that the AMNIOSENSE Blue pad can reliably rule in or rule out amniotic fluid leak as a cause of vaginal wetness in pregnancy, thus, can be adopted by hospitals as an amniotic fluid leak detection tool, and can be recommended by care providers for use in a home usage setting.

Study Group 1: Women attending the triage / delivery room with unidentified will be provided with an AMNIOSENSE Blue pad to use in hospital until they notice any wetness prior to a clinical assessment as per hospital standard procedure.

The clinician performing clinical diagnosis tests for amniotic fluid leak detection, according to the hospital standard procedure will be at all times blinded to the results of the AMNIOSENSE Blue pad.

Study Group 2: Women attending the obstetrical antenatal clinic for a routine antenatal visit > 36+0, and has not been referred for further assessment in triage/delivery unit by the physician will recruited to this study group (Study Group 2). Before leaving the antenatal clinic, they will be given one AMNIOSENSE Blue pad to use at home when vaginal wetness is experienced or in any case when they suspect that they have amniotic fluid leakage. The participant will be instructed to arrive at the hospital within 2 hours of applying the AMNIOSENSE Blue pad, regardless of the test results (positive or negative), to have a clinical diagnosis by the attending physician.

DETAILED DESCRIPTION:
This is a Prospective study to demonstrate that the AMNIOSENSE Blue pad can reliably rule in or rule out amniotic fluid leak as a cause of vaginal wetness in pregnancy, thus, can be adopted by hospitals as an amniotic fluid leak detection tool, and can be recommended by care providers for use in a home usage setting.

Study Group 1: Women attending the triage / delivery room with unidentified wetness will be provided with an AMNIOSENSE Blue pad to use in hospital until they notice any wetness but for no longer than 2 hours prior to a clinical assessment as per hospital standard procedure.

The clinician performing clinical diagnosis tests (clinical assessment) for amniotic fluid leak detection, according to the hospital standard procedure will be at all times blinded to the results of the AMNIOSENSE Blue pad.

Clinical diagnosis of ROM and subsequent management of care will be determined as per clinicians' judgment using the standard hospital procedures of ferning and/or positive Nitrazine testing and/or sterile speculum examination.

The research team or attending nurse (non-bias to the subject's result record) will read the results of the AMNIOSENSE Blue pad, record the results in the data collection forms, and place the AMNIOSENSE Blue pad in a sealed envelope labeled with the study ID. These results will not be communicated to the attending clinicians who will remain blinded.

In each case, the subject will also be required to read and record any occurrence of color change of the AMNIOSENSE Blue 10 minutes after removing the test on the designated form.

Study Group 2: Women attending the obstetrical antenatal clinic for a routine antenatal visit > 36+0, and has not been referred for further assessment in triage/delivery unit by the physician will recruited to this study group (Study Group 2). Before leaving the antenatal clinic, they will be given one AMNIOSENSE Blue pad to use at home when vaginal wetness is experienced or in any case when they suspect that they have amniotic fluid leakage.

The participants will be provided with instructions for use and also instructed to read the Instructions For Use (IFU) prior to applying the AMNIOSENSE Blue pad. They will be instructed to only apply the AMNIOSENSE Blue pad when they are planning to attend the triage/delivery unit for assessment of wetness/leaking. The participant will be instructed to arrive at the hospital within 2 hours of applying the AMNIOSENSE Blue pad, regardless of the test results (positive or negative), to have a clinical diagnosis by the attending physician.

Upon arrival to the triage/delivery unit, the participant and the attending nurse or research team member (non-bias to the subject's result record) will retrieve the AMNIOSENSE Blue pad and record the results in the designated data collection forms and place the AMNIOSENSE Blue pad in a sealed envelope labeled with the study ID. These results will not be communicated to the attending clinicians who will remain blinded.

In each case, the subject will also be required to read and record any occurrence of color change of the AMNIOSENSE Blue 10 minutes after removing the test on the designated form.

While in the hospital, participants will be managed according to standard hospital procedure at the discretion of the clinician and have clinical diagnostic tests (clinical assessment) for amniotic fluid leak detection, according to the hospital standard procedure. The clinician will be blinded to the results of the AMNIOSENSE Blue during the study, and as such subject treatment will be based only on the standard hospital diagnostic methods.

ELIGIBILITY:
Inclusion Criteria:

Group 1:

* Age 18 and above.
* Subject minimum 26+0 weeks of pregnancy.
* Subject presents with feeling of vaginal wetness.

Group 2:

* Age 18 and above
* Subject minimum 36+0 weeks of pregnancy
* Subject presents with a feeling of vaginal wetness, and has applied the AMNIOSENSE Blue pad prior to arriving at the triage/delivery unit

Exclusion Criteria:

* Subject is unable or unwilling to comply with study procedures
* Subject with active vaginal bleeding present at the time of admission to triage
* Evidence of a non-reassuring fetal status at the time of assessment in triage (abnormal fetal heart tracing)
* Subject has reported to have had sexual intercourse within the last 12 hours

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-07-01 (Estimated); Primary Completion 2017-12-30 (Estimated); Study Completion 2018-01-30 (Estimated)

PRIMARY OUTCOMES:
AmnioSense performance | 10 minutes
  The primary efficacy endpoints are: presence or absence of a blue or green stain on a yellow background as confirmed by the study team yielded by the AMNIOSENSE Blue, compared to the "hospital standard procedure" - final clinical diagnosis (positive/negative) to assess the agreement between the subject/study team reading and final clinical diagnosis, in both study group 1 (hospital usage and 2 home usage).

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Amanda, MD, Principal Investigator — Ottawa Hospital Research Institute

IPD SHARING:
Plan to Share IPD: No